CLINICAL TRIAL: NCT05950113
Title: Phase I Dose-Escalation Study of BCMA/CS1 Bispecific Chimeric Antigen Receptor (CAR)-T Cells for Relapsed/Refractory Multiple Myeloma
Brief Title: CART-BCMA/CS1 in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn before opening
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-000577; NCI-2023-04271 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Recurrent Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Biopsy; Cyclophosphamide; fludarabine; Fluorodeoxyglucose F18; Immunotherapy; Adjuvants, Immunologic; Leukapheresis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CART-BCMA/CS1) (Experimental): Patients undergo leukapheresis on 35 to 21 days before Infusion Day (I-Day -35 to I-Day -21) and receive cyclophosphamide IV over 60 minutes and fludarabine IV over 30 minutes on I-Days -5, -4, and -3. Patients then receive CART-BCMA/CS1 IV on I-Day-0 on study. Patients undergo ECHO, ECG and MRI during screening. Patients undergo bone marrow biopsy and/or bone marrow aspirate screening, between I-Day -28 to I-Day -5, I-Day 30, and at 1 year post CART-BCMA/CS1 infusion. Patients also undergo FDG PET/CT during screening, between I-Day -28 to I-Day -5, I-Day 90 and I-Day 180 and every 3 months thereafter.
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Procedure: Echocardiography; Drug: Fludarabine; Other: Fludeoxyglucose F-18; Other: Immunotherapy; Procedure: Leukapheresis; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Receive IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Fludarabine — Receive IV
  Other Names: Fluradosa
Other: Fludeoxyglucose F-18 — Receive IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Immunotherapy — Receive CART-BCMA/CS1 cells IV
  Other Names: Immunological; Immunological Therapy; Immunologically Directed Therapy
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase I trial studies the side effects and how well CART-BCMA/CS1 works in treating patients with multiple myeloma (MM) that has come back (relapsed) or that does not respond to treatment (refractory). Chimeric antigen receptor (CAR) T-cell therapy is a type of treatment in which a patient's T cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T cells are grown in the laboratory and given to the patient by infusion for treatment of certain cancers, including MM. Immune cells can be engineered to kill MM cells by inserting a piece of deoxyribonucleic acid (DNA) into the immune cells using a lentiviral vector, that allows them to recognize MM cells.

CART-BCMA cells are such modified T cells that target markers called CS1 or B-cell maturation antigen (BCMA), which is expressed by a type of white blood cell called a "B-cell", which are cells that may help the MM cells grow. These engineered CART-BCMA/CS1 cells may kill MM cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of CART-BCMA/CS1 cells in patients with R/R MM for determination of a recommended phase 2 dose (RP2D).

SECONDARY OBJECTIVES:

I. To describe the overall adverse event profile of CART-BCMA/CS1 cells. II. To investigate the efficacy of CART-BCMA/CS1 cells. III. To evaluate the persistence of CART-BCMA/CS1 cells.

EXPLORATORY OBJECTIVES:

I. To characterize the cytokine environment following CART-BCMA/CS1 cell infusion and to evaluate changes in the setting of CRS.

II. To evaluate changes in T-cell subsets and function following CART-BCMA/CS1 cell infusion.

III. To examine the change in expression of BCMA and CS1 on clonal plasma cells in the bone marrow and/or extramedullary disease after CART-BCMA/CS1 cell treatment.

IV. To evaluate for plasma-cell aplasia.

OUTLINE: This is a first-in-human, phase I, single-arm, open-label, dose-escalation study.

Patients undergo leukapheresis 35 to 21 days before Infusion Day (I-Day -35 to I-Day -21) and receive cyclophosphamide intravenously (IV) over 60 minutes and fludarabine IV over 30 minutes on I-Days -5, -4, and -3. Patients then receive the CART-BCMA/CS1 infusion IV on I-Day -0 on study. Patients undergo echocardiography (ECHO), electrocardiogram (ECG), and magnetic resonance imaging (MRI) during screening. Patients undergo bone marrow biopsy and/or bone marrow aspirate screening, between I-Day -28 to I-Day -5, I-Day 30, and at 1 year post CART-BCMA/CS1 infusion. Patients also undergo fluorodeoxyglucose F-18 (FDG) positron emission tomography/computed tomography (PET/CT) during screening, between I-Day -28 to I-Day -5, I-Day 90 and I-Day 180 and every 3 months thereafter.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months until 5 years, then annually for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma relapsed or refractory after at least three prior lines of therapy, including:

  * A proteasome inhibitor and immunomodulatory agent either alone or in combination
  * Anti-CD38 (Cluster of Differentiation 38) directed therapy
  * Patients previously treated with anti-BCMA directed therapy are allowed onto the study. Patients must not have a history of grade > 3 CRS or grade >= 3 immune effector cell associated neurotoxicity (ICANS) with prior anti-BCMA therapy
* Patients must have measurable MM as defined by at least one of the criteria below:

  * Serum M-protein >= 0.5 g/dl (5 g/L)
  * Urine M-protein >= 200 mg/24 h
  * Serum free light chain (FLC) assay: involved FLC level >= 10 mg/dl (100 mg/l) provided serum FLC ratio is abnormal
  * A biopsy-proven plasmacytoma
* Age >= 18 years old and =< 74 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1 x 10^9 cells/L. Granulocyte colony stimulating factor is permitted (within 30 days prior to enrollment using standard phase I criteria for organ function)
* Platelets >= 50 x 10^9/L. Without transfusion, growth factors may be used to achieve eligibility criteria (within 30 days prior to enrollment using standard phase I criteria for organ function)
* Hemoglobin >= 8 g/dL (with or without transfusion) (within 30 days prior to enrollment using standard phase I criteria for organ function)
* Aspartate and alanine aminotransferases (AST, ALT) =< 2.5 x upper limit of normal (ULN) (within 30 days prior to enrollment using standard phase I criteria for organ function)
* Total bilirubin =< 2 x ULN (except patients with documented Gilbert's syndrome) (Within 30 days prior to enrollment using standard phase I criteria for organ function)
* Creatinine clearance >= 30 mL/min (within 30 days prior to enrollment using standard phase I criteria for organ function)
* Must be willing and able to accept at least one leukapheresis procedure
* Must be willing and able to provide written informed consent

Exclusion Criteria:

* Inability to purify >= 5 x 10^8 CD62L-enriched cells from leukapheresis product
* Previously known hypersensitivity to any of the agents used in this study; known sensitivity to cyclophosphamide or fludarabine
* Received systemic treatment for multiple myeloma, including immunotherapy, within 14 days prior to initiation of lymphodepletion chemotherapy administration within this protocol. Consistent with current trials, patients may otherwise be given bridging therapy at the discretion of the lead study investigator
* Prior allogeneic hematopoietic stem cell transplantation
* Autologous hematopoietic stem cell transplantation within 12 weeks prior to enrollment. Patients who have received an autologous transplant over 12 weeks from enrollment will not be excluded and may participate in the trial
* Potential requirement for systemic corticosteroids or concurrent immunosuppressive drugs based on prior history or having received systemic steroids within the last 2 weeks prior to enrollment (inhaled or topical steroids at standard doses are allowed)
* Human immunodeficiency virus (HIV) seropositivity or other congenital or acquired immune deficiency state, which would increase the risk of opportunistic infections and other complications during chemotherapy-induced lymphodepletion. If there is a positive result in the infectious disease testing that was not previously known, the patient will be referred to their primary physician and/or infectious disease specialist
* Hepatitis B or C seropositivity with evidence of ongoing liver damage, which would increase the likelihood of hepatic toxicities from the lymphodepletion chemotherapy regimen and supportive treatments. Patients with hepatitis C seropositive disease but undetectable hepatic C virus (HCV) ribonucleic acid (RNA) viral load will be allowed in the trial. Patients with B seropositivity on antiviral therapy will be allowed in the trial
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol
* Known clinically active central nervous system involvement (CNS). Prior evidence of CNS involvement successfully treated will not be an exclusion for participation as long as they are deemed under control at the time of study enrollment and there are no neurological signs of potential CNS involvement. A brain magnetic resonance imaging (MRI) scan taken within 8 weeks of lymphodepletion may be used, otherwise a brain MRI must be performed to confirm absence of CNS involvement
* Oxygen saturation of =< 92% on room air
* A left ventricular ejection fraction =< 45%
* Pregnancy or breast-feeding. Female patients must be surgically sterile or be postmenopausal for two years or must agree to use effective contraception during the period of treatment and for 6 months afterwards. All female patients with reproductive potential must have a negative pregnancy test (serum/urine) at screening and again within 14 days from starting the lymphodepletion chemotherapy. The definition of effective contraception will be based on the judgment of the study investigators. Patients who are breastfeeding are not allowed on this study
* History of other malignancy in the past 3 years with the following exceptions:

  * Malignancy treated with curative intent and no known active disease
  * Adequately treated non-melanoma skin cancer without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductile carcinoma without evidence of disease
  * Prostate cancer with a Gleason score less than 6 with undetectable prostate specific antigen over 12 months
  * Adequately treated urothelial non-invasive carcinoma or carcinoma in situ
  * Similar neoplastic conditions with an expectation of greater than 95% disease free survival

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2027-03-28 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Within 28 days from CART-BCMA/CS1 cell infusion
  Will be assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v. 5). For cytokine release syndrome (CRS) and neurotoxicity, patients will be evaluated using the grading criteria outlined by the American Society for Transplantation and Cellular Therapy (ASTCT).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 15 years
  Will be assessed by CTCAE v. 5 and occurrence and grade of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) per ASTCT criteria.
Clinical response rate | Up to 2 years
  Will be assessed according to to the International Myeloma Working Group (IMWG) Uniform Response criteria, including minimum residual disease (MRD). MRD status for patients in complete remission (CR) will be summarized. Rates of best response of >= complete response (CR) or >= very good partial response (VGPR) may be summarized.
Overall response rate | Up to 2 years
  Will be summarized with the frequency count and percentage of patients in each category
Duration of response | Up to 2 years
  Will be measured after treatment from the time measurement criteria is met for stringent complete response (sCR), CR, VGPR, or partial response (PR) until the first date that progressive disease (PD) is objectively documented or until death. Will be summarized using the Kaplan-Meier method.
Overall survival | The date of CART-BCMA/CS1 cell infusion in the study until death, assessed up to 15 years
  Will be summarized using the Kaplan-Meier method. The Kaplan-Meier estimates for the 1-year Overall Survival (OS) rates and the 2-sided 95% confidence interval of the rates using the Greenwood's formula will be reported and will be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum) and will be summarized descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Progression free survival | The date of CART-BCMA/CS1 cell infusion until documentation of PD, or death due to any cause, assessed up to 2 years
  Will be summarized using the Kaplan-Meier method.
CART-BCMA/CS1 cell persistence | Up to 5 years
  Expansion and persistence of CART-BCMA/CS1 cells will be monitored with Real-time polymerase chain reaction (qPCR) specific to CART-BCMA/CS1 lentiviral elements in order to quantify the vector copy number. DNA will be extracted from peripheral blood cells and assessed with primers specific to genetic elements inserted by the lentivirus. Analysis will be performed to determine the number of days until CART-BCMA/CS1 cells are no longer detectable by polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Larson, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- Melanie Ayala Ceja, Los Angeles, California, United States